CLINICAL TRIAL: NCT06181708
Title: Estimating & Comparing the Performance, Clinical Effectiveness, and Cost-effectiveness of Current Diagnostic Options for Patients That Present to Primary Care With Suspected Venous Ulcers
Brief Title: Diagnostics in the Leg Ulcer Pathway
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23CX8458
Record Dates: First submitted 2023-11-10; First posted 2023-12-26 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary care practitioners: A one off questionnaire to be sent to primary care practitioners via qualtrics to determine the current practice in primary care for venous leg ulcer management and availability of services to onward referral.
  Interventions: Other: N/A - Questionnaire based study
- Vascular Scientists: A Delphi Consensus questionnaire will be performed via Qualtrics to determine the current practice for diagnosis and management of suspected venous leg ulcers in vascular scientist departments across the UK
  Interventions: Other: N/A - Questionnaire based study

INTERVENTIONS:
Other: N/A - Questionnaire based study — Questionnaire based study

SUMMARY:
This project aims to investigate 'The minimum diagnostic requirements for patients presenting to primary care with suspected venous ulcers.' In order to do this, the investigators intend to run a series of questionnaires with primary care services, vascular science services, and perform some cost effectiveness modelling on running diagnostic services in primary care and in secondary care settings. A one off questionnaire, designed in Qualtrics, will be sent out to primary care practitioners via social media and email contacts. This will be aimed at establishing their current role and any guidelines they follow with regards to the diagnosis and management of venous leg ulcers in primary care, and to determine their opinion of what this patient pathway should involve. A Delphi consensus will be carried out amongst vascular scientists across the UK to determine current and streamline future practice in diagnostics for patients with venous leg ulcers. The consensus will be achieved when there is ≥ 70% agreement. Cost effectiveness modelling will be carried out on two different scenarios of managing this cohort of patients, one in primary care and one in secondary care settings. Descriptive statistics will be performed on the results.

DETAILED DESCRIPTION:
The main objective of this project is to determine the role/position of diagnostic imaging in the patient journey for a patient with active or healed ulceration.

1. To determine the current practice in primary care for venous leg ulcer management and availability of services to onward referral.
2. To determine the current practice for diagnosis and management of suspected venous leg ulcers in vascular scientist departments across the UK
3. To establish what the minimum diagnostics should be for this cohort of patients including what scans should be performed and can a set criterion be applied to this cohort of patients.
4. To determine the cost effectiveness of implementing this in both primary and secondary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practitioners working in the UK will be recruited for the primary care questionnaire.
* Vascular Scientists working in a secondary care hospital in the UK will be recruited for the online delphi consensus.

Exclusion Criteria:

* Participants not meeting the inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care practitioners working in the UK and Vascular Scientists working in a secondary care hospital in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2025-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Care Practitioners | Vascular Scientists
Started | 92 | 43
Completed | 92 | 36
Not Completed | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Practitioners | Vascular Scientists | Total
Number analyzed (Participants) | 92 | 43 | 135
Age, Customized [Number; unit: years] — Age of participants not collected for this study. Population: Age of participant not collected for this study.
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of participants not collected for this study. Population: Gender of participants not collected for this study.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Primary Care Practitioners and the Management of Venous Leg Ulcers.
Description: What percentage of respondents have access to onward specialist referral for venous leg ulcer management? What percentage of primary care practitioners have access to refer for venous duplex imaging? What percentage of primary care practitioners felt there needs to be clearer guidelines on the management of patients with venous leg ulcers.
Time Frame: 3 months
Population: The overall response rate was 92, but it was not compulsory to answer every question in the questionnaire, so some questions had different response rates.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Practitioners
Number analyzed (Participants) | 92
Participants
  What % of respondents have access to onward specialist referral for venous leg ulcer management?: number analyzed (Participants) | 79
  What % of respondents have access to onward specialist referral for venous leg ulcer management? | 50
  What percentage of primary care practitioners have access to refer for venous duplex imaging?: number analyzed (Participants) | 75
  What percentage of primary care practitioners have access to refer for venous duplex imaging? | 34
  What % of PCP felt there needs to be clearer guidelines on management of patients with VLUs.: number analyzed (Participants) | 74
  What % of PCP felt there needs to be clearer guidelines on management of patients with VLUs. | 45

2. Primary Outcome: Vascular Scientists
Description: To determine a consensus on the diagnostic management of suspected venous leg ulcers in vascular scientist departments across the UK.
  What % of respondents felt there needed to be clearer guidelines on how to best manage these patients diagnostically? What % of respondents felt that specialist leg ulcer clinics should be run? What % felt patients should be able to access an ABPI as part of this clinic? What % felt patients should be able to access a venous duplex scan as part of this clinic? What % felt leg ulcer clinics should be held in secondary
Time Frame: 3 months
Population: There were 43 responses to the Delphi.
Measure: Count of Participants; unit: Participants
Arm/Group | Vascular Scientists
Number analyzed (Participants) | 43
Participants
  What % of respondents felt there needed to be clearer diagnostic guidelines?: number analyzed (Participants) | 39
  What % of respondents felt there needed to be clearer diagnostic guidelines? | 29
  What % of respondents felt that specialist leg ulcer clinics should be run?: number analyzed (Participants) | 36
  What % of respondents felt that specialist leg ulcer clinics should be run? | 33
  What % felt patients should be able to access an ABPI as part of this clinic?: number analyzed (Participants) | 34
  What % felt patients should be able to access an ABPI as part of this clinic? | 32
  What % felt patients should be able to access a venous duplex scan as part of this clinic?: number analyzed (Participants) | 33
  What % felt patients should be able to access a venous duplex scan as part of this clinic? | 24
  What % felt leg ulcer clinics should be held in secondary care?: number analyzed (Participants) | 33
  What % felt leg ulcer clinics should be held in secondary care? | 22
  What % felt compression bandaging should be removed before a venous insufficiency scan?: number analyzed (Participants) | 36
  What % felt compression bandaging should be removed before a venous insufficiency scan? | 34

ADVERSE EVENTS:
Time Frame: N/A. Adverse Events were not monitored/assessed
Description: Adverse Events were not monitored/assessed
Groups:
- Primary Care Practitioners: A one off questionnaire to be sent to primary care practitioners via qualtrics to determine the current practice in primary care for venous leg ulcer management and availability of services to onward referral.
  N/A - Questionnaire based study: Questionnaire based study and therefore adverse Events were not monitored/assessed.
- Vascular Scientists: A Delphi Consensus questionnaire will be performed via Qualtrics to determine the current practice for diagnosis and management of suspected venous leg ulcers in vascular scientist departments across the UK
  N/A - Questionnaire based study: Questionnaire based study and therefore adverse Events were not monitored/assessed.
Arm/Group | Primary Care Practitioners | Vascular Scientists
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT06181708/Prot_000.pdf